CLINICAL TRIAL: NCT03824535
Title: 18F-FSPG PET/CT and Integrated Biomarkers for Early Lung Cancer Detection in Patients With Indeterminate Pulmonary Nodules
Brief Title: 18F-FSPG PET/CT in Diagnosing Early Lung Cancer in Patients With Lung Nodules
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andrei Iagaru (Other)
Collaborators: Canary Foundation (Other); Boston University (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Andrei Iagaru, Associate Professor of Radiology (Nuclear Medicine), Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-46607; NCI-2019-00177 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); LUN0106 (Other: Stanford Cancer Institute Palo Alto); IRB-46607 (Other: Stanford IRB)
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Cigarette Smoker; Current Smoker; Former Smoker; Multiple Pulmonary Nodules; Pulmonary Nodule
Keywords: Indeterminate lung nodule
MeSH Terms: conditions — Smoking Cessation; Multiple Pulmonary Nodules | interventions — Tomography, X-Ray Computed; Tomography; Fluorodeoxyglucose F18; 4-(3-fluoropropyl)glutamic acid; Positron-Emission Tomography; Positron Emission Tomography Computed Tomography; Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (18F-FSPG PET/CT, 18F-FDG PET/CT) (Experimental): Patients receive 18F-FSPG IV and, undergo a PET/CT scan over 30-60 minutes. Within 24 hours-14 days, patients receive 18F-FDG IV and undergo a second PET/CT scan over 30-60 minutes.
  Interventions: Diagnostic Test: Computed Tomography; Drug: Fludeoxyglucose F-18; Drug: Fluorine F 18 L-glutamate Derivative BAY94-9392; Diagnostic Test: Positron Emission Tomography (PET/CT)

INTERVENTIONS:
Diagnostic Test: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Drug: Fludeoxyglucose F-18 — Given IV
  Other Names: 18-FDG; FDG; fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Drug: Fluorine F 18 L-glutamate Derivative BAY94-9392 — Given IV
  Other Names: (S)-4-(3-18F-fluoropropyl)-L-glutamic Acid; 18F-FSPG; BAY94-9392
Diagnostic Test: Positron Emission Tomography (PET/CT) — Undergo PET/CT
  Other Names: Positron Emission Tomography/computer tomography; CT Scan; PET Scan; Positron Emission Tomography; medical imaging

SUMMARY:
This phase II trial studies how well 18F-FSPG positron emission tomography (PET)/computed tomography (CT) work in diagnosing early lung cancer in patients with indeterminate lung nodules. PET imaging with an imaging agent called 18F-FDG is often used in combination with a PET/CT scanner to evaluate cancers. Giving 18F-FSPG before a PET/CT scan may work better in helping researchers diagnose early lung cancer in patients with lung nodules.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Comparison of fluorine F 18 L-glutamate derivative BAY94-9392 (18F-FSPG) accumulation with fludeoxyglucose F-18 (18F-FDG) accumulation to assess whether (4S)-4-(3-18F-Fluoropropyl)-L-Glutamate (18F-FSPG)-PET is better at discriminating between benign and malignant nodules.

SECONDARY OBJECTIVES:

I. To develop and validate early lung cancer detection biomarkers that would directly impact the growing need to integrate imaging and non-invasive molecular diagnostics for indeterminate pulmonary nodules and allow physicians to avoid unnecessary invasive procedures in patients with benign lung disease.

OUTLINE:

Patients receive 18F-FSPG intravenously (IV) and, undergo a PET/CT scan over 30-60 minutes. Within 24 hours-14 days, patients receive 18F-FDG and undergo a second PET/CT scan over 30-60 minutes.

After completion of study, patients are followed up within 24-72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary nodule between the size of 7 to 30 mm. Subjects with multiple nodules may be eligible if the dominant nodule is 7 to 30 mm
* Undergoing standard of care 18F-FDG PET imaging (for indeterminate pulmonary nodule)
* Current or former cigarette smoker, with >= 20 pack years
* Documented informed consent

Exclusion Criteria:

* History or previous diagnosis of lung cancer
* Cancer diagnosis within the last 5 years
* Pregnant or nursing

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carina Mari Aparici, Principal Investigator — Stanford Cancer Institute Palo Alto
Locations (1):
- Stanford Cancer Institute Palo Alto, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic (18F-FSPG PET/CT, 18F-FDG PET/CT): Patients received 18F-FSPG IV and, underwent a PET/CT scan over 30-60 minutes. Within 24 hours-14 days, patients received 18F-FDG IV and underwent a second PET/CT scan over 30-60 minutes.
  Computed Tomography: Undergo PET/CT
  Fludeoxyglucose F-18: Given IV
  Fluorine F 18 L-glutamate Derivative BAY94-9392: Given IV
  Positron Emission Tomography: Undergo PET/CT
Period: Overall Study
Arm/Group | Diagnostic (18F-FSPG PET/CT, 18F-FDG PET/CT)
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (18F-FSPG PET/CT, 18F-FDG PET/CT)
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Performance Metrics (Sensitivity, Specificity, PPV, NPV, and Accuracy) of Ultrasonography and Capnography for Malignant Lung Nodules
Description: The diagnostic performance of ultrasonography and capnography in detecting malignant lung nodules was assessed using sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and accuracy. Sensitivity and specificity were calculated to determine the ability to correctly identify malignant and non-malignant nodules, respectively. Results were compared to a predefined threshold of 75%, with all percentages reported as proportions of the total number of nodules analyzed. Confidence intervals were calculated for each metric to ensure precision and reliability in the estimates.
Time Frame: Through study completion, an average of 2 years and 6 months
Population: One lesion per participant was evaluated; therefore, lesion and participant counts match 1:1.
Measure: Number (95% Confidence Interval); unit: percentage
Units Other Than Participants: Nodules
Groups:
- Diagnostic (18F-FSPG PET/CT); Diagnostic (18F-FDG PET/CT): Patients received 18F-FSPG IV and, underwent a PET/CT scan over 30-60 minutes. Within 24 hours-14 days, patients received 18F-FDG IV and underwent a second PET/CT scan over 30-60 minutes.
  Computed Tomography: Undergo PET/CT
  Fludeoxyglucose F-18: Given IV
  Fluorine F 18 L-glutamate Derivative BAY94-9392: Given IV
  Positron Emission Tomography: Undergo PET/CT
Arm/Group | Diagnostic (18F-FSPG PET/CT) | Diagnostic (18F-FDG PET/CT)
Number analyzed (Participants) | 15 | 15
Number analyzed (Nodules) | 15 | 15
percentage
  Sensitivity | 100 [100 to 100] | 70 [35 to 93]
  Specificity | 100 [40 to 100] | 100 [40 to 100]
  Positive Predictive Value (PPV) | 100 [100 to 100] | 100 [100 to 100]
  Negative Predictive Value (NPV) | 100 [100 to 100] | 57 [34 to 77]
  Accuracy | 100 [77 to 100] | 79 [49 to 95]
Statistical Analysis 1: Comparison: Diagnostic (18F-FSPG PET/CT) vs Diagnostic (18F-FDG PET/CT); Analysis applies to the row 'Specificity' in the Outcome Measure data table; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was set at p < 0.05

2. Secondary Outcome: Improvement in Predictive Accuracy of Lung Nodule Diagnosis Using the C Statistic (Area Under the Curve, AUC)
Description: The predictive accuracy of the lung nodule diagnosis model was assessed using the C statistic, also referred to as the area under the receiver operating characteristic (ROC) curve (AUC). Improved performance was defined as a statistically significant increase (p < 0.05) in the C statistic, determined using the DeLong test for comparing correlated ROC curves. The Mann-Whitney U test was also used to compare the distributions of the C statistic between diagnostic methods. Results are reported as the mean C statistic with 95% confidence intervals for each diagnostic method.
Time Frame: Through study completion, an average of 2 years and 6 months
Measure: Mean (Standard Error); unit: probability
Units Other Than Participants: Nodules
Groups:
- Baseline Diagnostic (18F-FSPG PET/CT); Improved Diagnostic (18F-FDG PET/CT): Patients received 18F-FSPG IV and, underwent a PET/CT scan over 30-60 minutes. Within 24 hours-14 days, patients received 18F-FDG IV and underwent a second PET/CT scan over 30-60 minutes.
  Computed Tomography: Undergo PET/CT
  Fludeoxyglucose F-18: Given IV
  Fluorine F 18 L-glutamate Derivative BAY94-9392: Given IV
  Positron Emission Tomography: Undergo PET/CT
Arm/Group | Baseline Diagnostic (18F-FSPG PET/CT) | Improved Diagnostic (18F-FDG PET/CT)
Number analyzed (Participants) | 15 | 15
Number analyzed (Nodules) | 15 | 15
probability | 0.84 (0.1) | 1.0 (0.0)
Statistical Analysis 1: Comparison: Baseline Diagnostic (18F-FSPG PET/CT) vs Improved Diagnostic (18F-FDG PET/CT); Test type: Superiority; p = 0.004, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was predefined as p < 0.05
Statistical Analysis 2: Comparison: Baseline Diagnostic (18F-FSPG PET/CT) vs Improved Diagnostic (18F-FDG PET/CT); Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was predefined as p ≤ 0.05
Statistical Analysis 3: Comparison: Baseline Diagnostic (18F-FSPG PET/CT) vs Improved Diagnostic (18F-FDG PET/CT); Test type: Superiority; p = 0.06, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was predefined as p < 0.05

ADVERSE EVENTS:
Time Frame: Within 24 to 72hours after the 18F-FSPG PET/CT
Arm/Group | Diagnostic (18F-FSPG PET/CT, 18F-FDG PET/CT)
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/35/NCT03824535/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-24): https://cdn.clinicaltrials.gov/large-docs/35/NCT03824535/ICF_002.pdf